CLINICAL TRIAL: NCT00483262
Title: Phase I/II Trial of Combination CCI-779 (Temsirolimus) and Bortezomib (Velcade) in Relapsed and/or Relapsed/Refractory Multiple Myeloma
Brief Title: Combination CCI-779 (Temsirolimus) and Bortezomib (Velcade) in Relapsed and/or Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-365
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Results first posted 2013-05-10 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-10

CONDITIONS: Multiple Myeloma
Keywords: Temsirolimus; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — temsirolimus; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CCI779 and Bortezomib Phase I/II (Experimental): In Phase I part, 15 or 25 mg temsirolimus (CCI-779)and 1·3 or 1·6 mg/m² bortezomib was given once a week.In Phase II, patients received intravenous temsirolimus once a week on days 1, 8, 15, 22, and 29 for a cycle of 35 days, and intravenous bortezomib once a week on days 1, 8, 15, and 22 for a cycle of 35 days, the MTD ascertained in the Phase I part.
  Interventions: Drug: CCI-779; Drug: Bortezomib

INTERVENTIONS:
Drug: CCI-779 — Given by injection once a week for 5 weeks (5 weeks equals one cycle) for up to 8 cycles
  Other Names: Temsirolimus
Drug: Bortezomib — Given by injection once a week for 4 weeks (a cycle equals 5 weeks) for up to 8 cycles
  Other Names: Velcade

SUMMARY:
The purpose of this research study is to determine the safety of CCI-779 (Temsirolimus) and bortezomib (Velcade), and the highest dose of this drug that can be given to people safely. We will also be looking at how the combination of the two drugs may work against multiple myeloma. CCI-779 (Temsirolimus) is a drug that appears to stop myeloma cells from growing.

DETAILED DESCRIPTION:
* Since we are looking for the highest dose of CCI-779 (Temsirolimus) given in combination with bortezomib (Velcade) that can be given to people without causing the most serious or unmanageable side effects, not everyone who participates in this study will be receiving the same amount of either drug.
* During the study treatment, participants will be given some medications to decrease the chance they they will have an allergic reaction to CCI-779 (Temsirolimus). After these drugs are given, participants will be receive bortezomib (Velcade) by injection followed by an injection of CCI-779 (Temsirolimus). These drugs wil be given once a week for four weeks (on Days 1, 8, 15, and 22). On the fifth week (Day 29), participants will be given only CCI-779 along with the drugs to decrease the chance of an allergic reaction.
* The cycle will last 35 days and will occur twice before the doctor evaluates for response. The cycles will be repeated for up to 8 cycles as long as the participant does not have any severe or unmanageable side effects and the disease is responding to treatment.
* While receiving study treatment, participants will be seen at the clinic at the start of each cycle for the following: complete physical examination, blood work, urine collection, x-ray of bones (if study doctor deems necessary) and an electrocardiogram (prior to treatment and at the end of treatment)
* A bone skeletal survey will be performed at the end of treatment to measure the size of the participants tumors.
* After 8 cycles of treatment or if the participant has ended treatment, more tests will be performed. A physical exam, blood work, urine collection, skeletal survey, electrocardiogram, bone marrow biopsy and aspirate will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must have received prior therapy for their myeloma and have relapsed and/or relapsed/refractory multiple myeloma
* Monoclonal protein in the serum of greater than or equal to 1 gm/dL or monoclonal light chain in the urine protein electrophoresis of greater than or equal to 200mg/24 hours, or measurable light chains by free light chain assay of greater than or equal to 10mg/dl, or measurable plasmacytoma
* ECOG Performance Status 0, 1 or 2
* Laboratory values as outlined in the protocol

Exclusion Criteria:

* Uncontrolled infection
* Cytotoxic chemotherapy less than 2 weeks, or biologic therapy less than 2 weeks, or corticosteroids less than 2 weeks prior to registration. Patients may be receiving chronic corticosteroids if they are being given for disorders other than myeloma.
* Pregnant or nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational within 14 days before enrollment
* Known to be HIV positive
* Myocardial infarction within 6 months prior to enrollment or has NYHA Class III or IV hear failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Hypersensitivity to bortezomib, boron or mannitol
* Serious medical or psychiatric illness likely to interfere with participation in this clinical trial
* Patients who may need or are receiving live vaccines for immunization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-05; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in Saint Louis, St Louis, Missouri

REFERENCES:
- [Result] Ghobrial IM, Weller E, Vij R, Munshi NC, Banwait R, Bagshaw M, Schlossman R, Leduc R, Chuma S, Kunsman J, Laubach J, Jakubowiak AJ, Maiso P, Roccaro A, Armand P, Dollard A, Warren D, Harris B, Poon T, Sam A, Rodig S, Anderson KC, Richardson PG. Weekly bortezomib in combination with temsirolimus in relapsed or relapsed and refractory multiple myeloma: a multicentre, phase 1/2, open-label, dose-escalation study. Lancet Oncol. 2011 Mar;12(3):263-72. doi: 10.1016/S1470-2045(11)70028-6. Epub 2011 Feb 21. PMID 21345726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June, 2007, and December, 2009, we enrolled patients into our open-label, dose-escalation study at three centres in the USA (Dana-Farber Cancer Institute, Boston, MA; Washington University, St Louis, MO; and the University of Michigan, Ann Arbor, MI).
Groups:
- CCI779 and Bortezomib Phase I: CCI779 and Bortezomib, Phase I part of this Phase I/II study
- CCI779 and Bortezomib Phase II: CCI779 and Bortezomib, Phase II part of this Phase I/II study
Period: Overall Study
Arm/Group | CCI779 and Bortezomib Phase I | CCI779 and Bortezomib Phase II
Started | 20 | 43
Completed | 20 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CCI779 and Bortezomib Phase I: CCI779 and Bortezomib Phase I part of this Phase I/II study.
- CCI779 and Bortezomib Phase II: CCI779 and Bortezomib Phase II part of this Phase I/II study
- Total: Total of all reporting groups
Arm/Group | CCI779 and Bortezomib Phase I | CCI779 and Bortezomib Phase II | Total
Number analyzed (Participants) | 20 | 43 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 23 | 38
  >=65 years | 5 | 20 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 24 | 31
  Male | 13 | 19 | 32
Region of Enrollment [Number; unit: participants]
  United States | 20 | 43 | 63

OUTCOME MEASURES:

1. Primary Outcome: Toxicity. Number of Patients With Specific Toxicities Are Reported.
Description: Toxicity of CCI-779 (Temsirolimus) and bortezomib (Velcade) in patients with multiple myeloma.
Time Frame: 10 months
Population: Any patient who was treated was included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- CCI779 Toxicity Phase I: Toxicity of CCI779 and velcade in the phase I part of this phase I/II study. CTC criteria used.
- CCI779 Toxicity Phase II: Toxicity of CCI779 and velcade in the phase II part of this phase I/II study. CTC criteria used
Arm/Group | CCI779 Toxicity Phase I | CCI779 Toxicity Phase II
Number analyzed (Participants) | 20 | 43
percentage of patients | 90 [72 to 98] | 79 [66 to 89]
Statistical Analysis 1: Comparison: CCI779 Toxicity Phase I; Single Arm Study; Test type: Superiority or Other; >= grade 3 adverse event proportion = .90, 90% CI 2-sided [.72 to .98] — Estimated proportion of patients with a adverse event of grade 3 or higher
Statistical Analysis 2: Comparison: CCI779 Toxicity Phase II; Phase II toxicity; Test type: Superiority or Other; toxicity grade >=3 proportion = .79, 90% CI 2-sided [.66 to .89] — No comparison. Estimate the proportion of patients with grade 3 or higher toxicity

2. Primary Outcome: Best Response to Combination Treatment
Description: Response rate of PR or better to the combination treatment of CCI-779 (Temsirolimus) and bortezomib (Velcade) in patients with relapsed or refractory multiple myeloma
Time Frame: 10 months
Population: All patients included in analysis
Measure: Number (90% Confidence Interval); unit: percentage of patients
Groups:
- CCI779 Response Phase I: Response of PR or better per the Blade criteria in phase I part of this phase I/II study of CCI779 and velcade
- CCI779 Response Phase II: Response of PR or better per the Blade criteria in phase II part of this phase I/II study of CCI779 and velcade
Arm/Group | CCI779 Response Phase I | CCI779 Response Phase II
Number analyzed (Participants) | 20 | 43
percentage of patients | 10 [2 to 28] | 33 [21 to 47]
Statistical Analysis 1: Comparison: CCI779 Response Phase I; Phase I part of this phase I/II study; Test type: Superiority or Other; response rate of PR or better = 0.10, 90% CI 2-sided [.02 to .28] — Response of PR or better
Statistical Analysis 2: Comparison: CCI779 Response Phase II; Phase II part of this phase I/II study; Test type: Superiority or Other; response rate of PR or better = 0.33, 90% CI 2-sided [0.21 to 0.47] — Response of PR or better

3. Secondary Outcome: Progression-Free Survival
Description: Median time to progression or death
Time Frame: 10 months
Measure: Median (95% Confidence Interval); unit: month
Groups:
- CCI779 PFS Phase I: Progression-free survival results from the phase I part of the phase I/II CCI779 with velcade study.
- CCI779 PFS Phase II: Progression-free survival results from the phase II part of the phase I/II CCI779 with velcade study.
Arm/Group | CCI779 PFS Phase I | CCI779 PFS Phase II
Number analyzed (Participants) | 20 | 43
month | 5.7 [1.5 to 9.2] | 5.0 [3.9 to 6.4]

ADVERSE EVENTS:
Time Frame: June 2007 to December 2009
Groups:
- Adverse Events CCI779 and Bortezomib Phase I: Adverse Events of CCI779 and Bortezomib in the phase I part of this phase I/II study.
- Adverse Events CCI779 and Bortezomib Phase II: Adverse Events of CCI779 and Bortezomib in Phase II part of this Phase I/II study.
Arm/Group | Adverse Events CCI779 and Bortezomib Phase I | Adverse Events CCI779 and Bortezomib Phase II
Serious Adverse Events (participants affected / at risk) | 13/20 | 25/43
Other Adverse Events (participants affected / at risk) | 18/20 | 34/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adverse Events CCI779 and Bortezomib Phase I (N=20) | Adverse Events CCI779 and Bortezomib Phase II (N=43)
Neutropenia (Blood and lymphatic system disorders) | 9 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 25
Leukopenia (Blood and lymphatic system disorders) | 7 | 10
Lymphopenia (Blood and lymphatic system disorders) | 10 | 24
Anemia (Blood and lymphatic system disorders) | 5 | 7
Diarrhea (Gastrointestinal disorders) | 0 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events CCI779 and Bortezomib Phase I (N=20) | Adverse Events CCI779 and Bortezomib Phase II (N=43)
Thromobocytopenia (Blood and lymphatic system disorders) | 13 (19) | 34 (36)
Neutropenia (Blood and lymphatic system disorders) | 18 (18) | 25 (27)
Leucopenia (Blood and lymphatic system disorders) | 14 (14) | 30 (32)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 13 (13) | 14 (14)
Anaemia (Blood and lymphatic system disorders) | 11 (12) | 25 (25)
Diarrhea (Gastrointestinal disorders) | 11 (11) | 22 (22)
Fatigue (General disorders) | 11 (11) | 21 (21)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (10) | 12 (12)
Lymphopenia (Blood and lymphatic system disorders) | 10 (10) | 25 (26)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 (7) | 11 (11)
Nausea (Gastrointestinal disorders) | 5 (6) | 15 (15)
Anorexia (Gastrointestinal disorders) | 5 (5) | 10 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 5 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (6)
Vomiting (Gastrointestinal disorders) | 1 (2) | 11 (11)
Weight loss (General disorders) | 2 (2) | 0 (0)
Herpes-Zoster infection (Infections and infestations) | 2 (2) | 2 (2)
Cardiac ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Blood infection with grade 0-2 neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Mucositis/stomatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neuropathy (sensory) (Nervous system disorders) | 0 (0) | 11 (11)
Neuropathy (motor) (Nervous system disorders) | 0 (0) | 7 (7)
Nose, haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 7 (7)
Abdomen, pain (General disorders) | 0 (0) | 4 (4)
Colitis, infectious (Infections and infestations) | 0 (0) | 2 (2)
Haemorrhage (lung and rectum) (General disorders) | 0 (0) | 3 (3)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Necrosis and obstruction, small bowel (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes